CLINICAL TRIAL: NCT00004847
Title: Diagnosis, Pathophysiology, and Molecular Biology of Pheochromocytoma and Paraganglioma
Brief Title: Diagnosis of Pheochromocytoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 000093; 00-CH-0093
Record Dates: First submitted 2000-03-02; First posted 2000-03-03 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-09-23

CONDITIONS: Pheochromocytoma; Endocrine Disease; Endocrine Diseases
Keywords: Genetics; Metanephrines; PET; Catecholamines
MeSH Terms: conditions — Pheochromocytoma; Endocrine System Diseases | interventions — fluorodopa F 18; 6-fluorodopamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adults or children with suspected PHEO/PGL (Experimental): Patients are adults or children of any age with known, sporadic or familial PHEO/PGL
  Interventions: Drug: ([18F]-DOPA); Drug: ([18F]-6F-DA)

INTERVENTIONS:
Drug: ([18F]-DOPA) — is L 3, 4 dihydroxyphenylalanine (L-DOPA) labeled with the radioactive isotope 18F. In general, PPGLs belong to the group of neuroendocrine tumors. This heterogeneous group of tumors takes up amino acids, transforms them into biogenic amines (dopamine and serotonin) by decarboxylation and stores the amines in vesicles. L DOPA is a precursor of catecholamines (dopamine, norepinephrine and epinephrine). Epinephrine conversion to dopamine is catalyzed by the aromatic amino acid decarboxylase. According to previous and current studies, [18F]-DOPA PET is highly sensitive and specific for detection of PHEO/PGL67-69. However, there are only a few reports in the literature using [18F]-DOPA as a PET agent and particularly for patients with metastatic PPGLs. PET imaging will be done together with either a CT, an MRI or both modalities.
Drug: ([18F]-6F-DA) — is an imaging agent developed at the NIH, that may improve specificity and sensitivity in the localization of PPGLs. [18F]-6F-DA enters cells via the membrane norepinephrine transporter. Once inside cells, [18F]-6F-DA is translocated via the vesicular monoamine transporter into storage vesicles, where the radioactivity is concentrated. After injection of [18F]-6F-DA, the much faster disappearance of [18F]-6F-DA-derived radioactivity from the bloodstream and non-neuronal cells than from chromaffin cells should enable rapid visualization of PPGLs by PET scanning.

SUMMARY:
The goal of this study is to develop better methods of diagnosis, localization, and treatment for pheochromocytomas. These tumors, which usually arise from the adrenal glands, are often difficult to detect with current methods. Pheochromocytomas release chemicals called catecholamines, causing high blood pressure. Undetected, the tumors can lead to severe medical consequences, including stroke, heart attack and sudden death, in situations that would normally pose little or no risk, such as surgery, general anesthesia or childbirth.

Patients with pheochromocytoma may be eligible for this study. Candidates will be screened with a medical history and physical examination, electrocardiogram, and blood and urine tests. Study participants will undergo blood, urine, and imaging tests, described below, to detect pheochromocytoma. If a tumor is found, the patient will be offered surgery. If surgery is not feasible (for example, if there are multiple tumors that cannot be removed), evaluations will continue in follow-up visits. If the tumor cannot be found, the patient will be offered medical treatment and efforts to detect the tumor will continue. Main diagnostic and research tests may include the following:

1. Blood tests - mainly measurements of plasma or urine catecholamines and metanephrines as well as methoxytyramine. If necessary the clonidine suppression test can be carried out.
2. Standard imaging tests - Non-investigational imaging tests include computed tomography (CT), magnetic resonance imaging (MRI), sonography, and 123I-MIBG scintigraphy and FDG (positron emission tomography) PET/CT. These scans may be done before and/or after surgical removal of pheochromocytoma.
3. Research PET scanning is done using an injection of radioactive compounds. Patients may undergo 18F-FDOPA, 18F-DA, as well as 68Ga-DOTATATE PET/CT . Each scan takes up to about 2 hours.
4. Genetic testing - A small blood sample is collected for DNA analysis and other analyses.

DETAILED DESCRIPTION:
Pheochromocytomas (PHEOs) and paragangliomas (PGLs) are rare and clinically important chromaffin cell tumors that typically arise from the adrenal gland or from extra-adrenal paraganglia, respectively. The clinical features and consequences of PHEO/PGL result from the release of catecholamines (norepinephrine and/or epinephrine). An undetected PHEO/PGL poses a hazard to patients undergoing surgery, childbirth, or general anesthesia, due to the potential for excess catecholamine secretion, which can result in significant, often catastrophic outcomes. Diagnosing and localizing a PHEO/PGL can be challenging. Plasma and urinary catecholamines as well as their metabolites and radio-iodinated metaiodobenzylguanidine (MIBG) scanning can yield false-positive/negative results in patients harboring the tumor. Computed tomography (CT) and magnetic resonance imaging (MRI) lack sufficient specificity. The molecular mechanisms by which genotypic changes predispose to the development of PHEO/PGL remain unknown - even in patients with identified pathogenic variants. Moreover, in patients with hereditary predispositions, PHEOs/PGLs differ in terms of their growth, malignant potential, catecholamine phenotype, responses to standard screening tests, various imaging modalities and therefore subsequently, different therapeutic options. This protocol focuses on developmental, molecular, genetic, epigenetic, proteomic, metabolomics, immunologic and other types of studies to investigate the bases for predisposition to develop PHEOs/PGLs and for expression of different neurochemical and other phenotypes and malignant potentials including therapeutic responses. Furthermore, this protocol will also use new imaging approaches, for example [18F]-6F-dopamine ([18F]-6F-DA), and [18F]-L-3,4-dihydroxyphenylalanine ([18F]-FDOPA) positron emission tomography (PET)/CT, as well as dynamic contrast-enhanced MRI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients are eligible for inclusion in this study if they are adults or children of age 3 years old and up with known, sporadic or familial PHEO/PGL, on the basis of one or more of the following:

1. High levels of blood or urinary catecholamines, metanephrines, methoxytyramine or chromogranin A.
2. Highly suspected presence of PHEO/PGL based on imaging studies, even with normal biochemistry.
3. Personal or family history of PHEO/PGL or genetic pathogenic variants known to predispose individuals to develop PHEO/PGL.

Signed informed consent is required. The informed consent may be signed by the patient, parent/guardian in pediatric patients or legally authorized representative (LAR) in adults who lack-decision making capacity to consent to research participation.

Patients must have an outside general practitioner or endocrinologist. Patients with metastatic disease must also have an outside oncologist.

Family Members of Patients Arm (Linkage Analysis)

Participants are eligible for inclusion in this study arm if they are:

* Adult family members of patients enrolled in this study;
* The index family member in this study has a suspected hereditary PHEO/PGL based on previous genetic testing and other suspicious hereditory patterns such as family history of multiple individuals with PHEO/PGL; early age of disease onset; multiplicity of primary tumors; recurrence, etc. and
* Signed informed consent form is required

EXCLUSION CRITERIA:

Potential patients will be excluded on the basis of one or more of the following:

1. Pregnant or breastfeeding women
2. Severe cardiac dysfunction
3. Currently on dialysis

A pregnancy test is performed in women of childbearing age (up to age 55) as a screening after consenting. If a patient is found to have a positive pregnancy test, her participation in this protocol will be terminated. The patient can enroll or re-enroll in the protocol when she is no longer pregnant or breastfeeding.

In-person participating patients who are not willing to return to the NIH (e.g., after surgery or an initial evaluation) for more than 2 years may be removed from the protocol.

SPECIFIC INCLUSION/EXCLUSION CRITERIA FOR IMAGING STUDIES WITHIN OUR PROTOCOL:

In adult patients (Excludes Linkage Analysis Arm)

Imaging studies are not done in patients that have the following exclusion criteria:

* Inability to lie still for the entire imaging time (e.g., cough, severe arthritis, etc.).
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (e.g., severe claustrophobia, radiation phobia, etc.)
* Any additional medical conditions, serious illness, or other extenuating circumstance that, in the opinion of the Principal Investigator, may significantly interfere with study compliance.

In pediatric patients:

Inclusion criteria for research PET imaging in children:

* Children over 10 years old with very high suspicion of sporadic or familial PHEO/PGL based on at least one of the following:

  * The presence of new onset of symptoms typical of PHEO/PGL such as hypertension or hypertensive episodes, sweating, headaches, pallor, palpitations, drug resistant hypertension, etc.
  * Family history of PHEO/PGL or genetic pathogenic variants known to predispose individuals to develop these tumors.
  * The presence of a tumor on conventional imaging including ultrasound, CT and/or MRI or [123I]-MIBG or PET imaging not limited to [18F]-FDG.
* Children must give informed assent and be willing to return to the NIH for follow-up.

Exclusion criteria for research PET imaging in children:

* Children of less than 10 years of age.
* Children with impaired mental capacity that precludes informed assent.
* Inability to lie still for the entire imaging time (e.g., cough, turbulent children, severe claustrophobia, etc.).

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2000-03-22 (Actual); Primary Completion 2048-11-30 (Estimated); Study Completion 2048-11-30 (Estimated)

PRIMARY OUTCOMES:
To study specific genotypes, biochemical and imaging phenotypes of patients with various pheochromocytomas and paragangliomas.To stuty potential treatment options for metastatic pheochromocytoma and paraganglioma using cell cultures, cell ... | Baseline
  To study specific genotypes, biochemical and imaging phenotypes of patients with various pheochromocytomas and paragangliomas.To stuty potential treatment options for metastatic pheochromocytoma and paraganglioma using cell cultures, cell lines, animal

SECONDARY OUTCOMES:
To educate health care professionals and patients about pheochromocytoma and paraganglioma | end of study
  To educate health care professionals and patients about pheochromocytoma and paraganglioma

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Gordon, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Jha A, Patel M, Carrasquillo JA, Ling A, Millo C, Saboury B, Chen CC, Wakim P, Gonzales MK, Meuter L, Knue M, Talvacchio S, Herscovitch P, Rivero JD, Chen AP, Nilubol N, Taieb D, Lin FI, Civelek AC, Pacak K. Sporadic Primary Pheochromocytoma: A Prospective Intraindividual Comparison of Six Imaging Tests (CT, MRI, and PET/CT Using 68Ga-DOTATATE, FDG, 18F-FDOPA, and 18F-FDA). AJR Am J Roentgenol. 2022 Feb;218(2):342-350. doi: 10.2214/AJR.21.26071. Epub 2021 Aug 25. PMID 34431366
- [Derived] Wolf KI, Jha A, van Berkel A, Wild D, Janssen I, Millo CM, Janssen MJR, Gonzales MK, Timmers HJKM, Pacak K. Eruption of Metastatic Paraganglioma After Successful Therapy with 177Lu/90Y-DOTATOC and 177Lu-DOTATATE. Nucl Med Mol Imaging. 2019 Jun;53(3):223-230. doi: 10.1007/s13139-019-00579-w. Epub 2019 Feb 22. PMID 31231443
- [Derived] Abdul Sater Z, Jha A, Mandl A, Mangelen SK, Carrasquillo JA, Ling A, Gonzales MK, Lopes Abath Neto O, Miettinen M, Adams KT, Nockel P, El Lakis M, Pacak K. Gallbladder Paraganglioma Associated with SDHD Mutation: a Potential Pitfall on 18F-FDOPA PET Imaging. Nucl Med Mol Imaging. 2019 Apr;53(2):144-147. doi: 10.1007/s13139-018-0558-1. Epub 2019 Feb 19. PMID 31057686
- [Derived] Taieb D, Jha A, Guerin C, Pang Y, Adams KT, Chen CC, Romanet P, Roche P, Essamet W, Ling A, Quezado MM, Castinetti F, Sebag F, Pacak K. 18F-FDOPA PET/CT Imaging of MAX-Related Pheochromocytoma. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1574-1582. doi: 10.1210/jc.2017-02324. PMID 29534198
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-CH-0093.html